CLINICAL TRIAL: NCT07131475
Title: ReBlast Precision (Precision Biomarkers to Detect Brain Injury in Active-Duty United States Special Operations Forces With Repeated Blast Exposure)
Brief Title: Precision Biomarkers to Detect Brain Injury in Active-Duty United States Special Operations Forces With Repeated Blast Exposure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of South Florida (Other); Navy SEAL Foundation (Unknown); National Institutes of Health (NIH) (NIH); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025P000608; H9240525FE002 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2025-07-24; First posted 2025-08-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Blast Injury
Keywords: repeated blast exposure; Special Operations Forces; traumatic brain injury
MeSH Terms: conditions — Blast Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This diagnostic study of a single group - active-duty United States Navy SEALs -will utilize PBR28 TSPO PET. Use of the PBR tracer is overseen by the U.S. FDA. Thus, this study is considered "interventional". However, given that the purpose of the study is to develop an initial diagnostic testing protocol for repeated blast brain injury, the typical Phase criteria for therapeutic trials do not apply here. We have selected "Phase 2" from the required list of choices, because the safety of the PRB tracer has been previously established (hence Phase 1 is not appropriate) and because this is not a definitive efficacy study (hence Phase 3 is not appropriate).
Masking Description: The investigators analyzing the MRI, cognitive, psychological, physical symptom, and exposure data will be blinded to the PRB28 TSPO PET results. Similarly, the investigators analyzing the PBR28 TSPO PET results will be blinded to all other data elements. The participants will be also be blinded to PBR28 TSPO PET results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active-duty United States Navy SEALs (Experimental): All SEAL participants will undergo comprehensive, longitudinal assessments of their exposures, cognitive performance, psychological health, physical symptoms, neuroimaging biomarkers, and blood biomarkers.
  Interventions: Drug: PBR28 TSPO PET

INTERVENTIONS:
Drug: PBR28 TSPO PET — Each SEAL participant will undergo brain imaging with PBR28 translocator protein (TSPO) positron emission tomography (PET) at study enrollment and at 1-year follow up.

SUMMARY:
This is a 4-year, longitudinal study of 100 active-duty Navy SEALs. The goal of the study is to determine whether repeated blast exposure affects SEAL brain health and to develop an initial diagnostic testing protocol that detects repeated blast brain injury.

DETAILED DESCRIPTION:
Participants will travel to Massachusetts General Hospital (MGH) in Boston, MA for a 1-day study visit at enrollment (baseline) and 1-year follow-up. At each visit to MGH, participants will have brain scans, blood tests, and assessments of cognitive performance, psychological health, and physical symptoms. Every 3 months between the baseline and follow-up visits to Boston, there will be brief (~1 hour) assessments via phone or video teleconference.

ELIGIBILITY:
Inclusion Criteria:

1. Active-duty Navy SEAL Service Member
2. Early career SEAL (0-2 years) or mid-late career SEAL (10-15 years)
3. Age 18-50 years
4. Males, regardless of race or ethnicity

Exclusion Criteria:

1. History of moderate or severe TBI
2. History of major neurological disorder
3. Untreated or unstable severe psychiatric condition
4. Current severe medical condition that requires long-term treatment
5. Any condition that may cause undue risk to the participant or create a logistical contraindication
6. MRI contraindication
7. PET contraindication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
neuroimaging biomarkers | 1 year
  TSPO tracer uptake within the brain on TSPO PET, functional connectivity of the executive control, default and salience networks on resting-state functional MRI and diffusion MRI, and brain signal abnormalities on multidimensional MRI
blood biomarkers | 1 year
  tau, ptau, bd-tau, NF-L, GFAP, UCH-L1, IL-6, IL-10, TNF alpha
neuropsychiatric symptoms | 1 year
  Neurobehavioral Symptom Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
USSOCOM regulations prevent public release of the data generated for the current study. Future requests for these data may be submitted to the corresponding author and will then need to be vetted by USSOCOM.

REFERENCES:
- [Background] Gilmore N, Tseng CJ, Maffei C, Tromly SL, Deary KB, McKinney IR, Kelemen JN, Healy BC, Hu CG, Ramos-Llorden G, Masood M, Cali RJ, Guo J, Belanger HG, Yao EF, Baxter T, Fischl B, Foulkes AS, Polimeni JR, Rosen BR, Perl DP, Hooker JM, Zurcher NR, Huang SY, Kimberly WT, Greve DN, Mac Donald CL, Dams-O'Connor K, Bodien YG, Edlow BL. Impact of repeated blast exposure on active-duty United States Special Operations Forces. Proc Natl Acad Sci U S A. 2024 May 7;121(19):e2313568121. doi: 10.1073/pnas.2313568121. Epub 2024 Apr 22. PMID 38648470